CLINICAL TRIAL: NCT05571189
Title: Home Rehabilitation After Acute Pulmonary Embolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: American College of Chest Physicians (Other)
Responsible Party: Principal Investigator, Daniel Lachant, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00007680
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants who receive daily activity message (Experimental): The intervention group will receive instructions for a daily activity sent through SMS text message or email.
  Interventions: Behavioral: Daily Activity Text
- Participants who receive control message (Placebo Comparator): The control group will receive daily messages to help with blinding sent through text message or email. The messages will not include activity tasks and will include phrases such as "I hope you have a good day".
  Interventions: Behavioral: Control Text

INTERVENTIONS:
Behavioral: Daily Activity Text — Participants will receive a text each day with instructions about the daily activity they should complete for that day.
  Arms: Participants who receive daily activity message
Behavioral: Control Text — Participants will receive a text each day with no instructions about daily activity. It will have messages like "have a nice day."
  Arms: Participants who receive control message

SUMMARY:
The purpose of this study is to evaluate whether a home rehabilitation program after hospitalization for acute pulmonary embolism (PE) improves clinical outcomes at 3 months compared to usual care. Daily physical activity tasks that incorporate heart rate monitoring will be sent through email or text. This information could help improve the management of acute PE.

ELIGIBILITY:
Inclusion Criteria:

* English speaking (>18 years old). Daily messages will be sent in English.
* Acute PE with right ventricular enlargement or dysfunction defined by echocardiogram report, CT Angiogram report, or elevated cardiac biomarker (NT-pro BNP or troponin).
* Baseline testing started within 7 days of hospital discharge.

Exclusion Criteria:

* Pregnancy.
* Cardiac Effort >2.5 beats/m during 6MWT. This is for safety.
* Cardiac Effort <1.2 beats/m during 6MWT. They are unlikely to benefit.
* Resting tachycardia >120 beats/m during screening or at hospital discharge.
* Suspicion for Chronic Thromboembolic Pulmonary Hypertension.
* Systolic blood pressure >180 mmHg during screening or at hospital discharge.
* Inability to walk.
* Estimated prognosis <12 months at the time of discharge due to underlying co-morbidities.
* Advanced neurologic disease.
* Lack of access to email or text messaging.
* Inability to follow daily instructions.
* Participation in a structured exercise routine at least three days per week in the prior four weeks.
* Principal Investigator discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
mean change in vector magnitude count as measured by actigraphy | 10 weeks
  The Actigraph triaxial accelerometer will be used to monitor continuous activity at home on the non-dominant wrist. The accelerometer data will be downloaded and will include the vector magnitude count.
mean change in mean amplitude deviation as measured by actigraphy | 10 weeks
  The Actigraph triaxial accelerometer will be used to monitor continuous activity at home on the non-dominant wrist. The accelerometer data will be downloaded and will include the mean amplitude deviation.

SECONDARY OUTCOMES:
proportion of participants with post-PE syndrome | 12 weeks
  Participants will be evaluated by a physician to determine if they have post PE-syndrome
mean change in steps as measured by Actigraph | 12 weeks
  The Actigraph triaxial accelerometer will be used to monitor the number of steps taken at home on the non-dominant wrist. The accelerometer data will be downloaded and will include the step count.
mean change in activity as measured by Actigraph | 12 weeks
  The Actigraph triaxial accelerometer will be used to monitor the amount of activity taken at home on the non-dominant wrist. The accelerometer data will be downloaded and will include the amount of activity.
mean change in quality of life as measured by PROMIS | 12 weeks
  The PROMIS questionnaire ranges from 0-99 with higher scores indicating worse outcome.
mean change in quality of life as measured by Emphasis 10 | 12 weeks
  The Emphasis 10 questionnaire ranges from 0-50 with higher scores indicating worse quality of life.
mean change in quality of life as measured by Pulmonary Embolism quality of life questionnaire | 12 weeks
  The pulmonary embolism quality of life questionnaire ranges from 1 to 27 with higher scores indicating worse outcomes.
mean change in 6 minute walking distance | 12 weeks
mean change in heart rate during a 6 minute walk | 12 weeks
mean change in oxygen use during a 6 minute walk | 12 weeks
  Oxygen use will be measured by a measured by portable K5 metabolic analyzer.
mean change in carbon dioxide production during a 6 minute walk | 12 weeks
  Carbon Dioxide use will be measured by a measured by portable K5 metabolic analyzer.
proportion or subjects who develop chronic thromboembolic pulmonary hypertension | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lachant, DO, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No